CLINICAL TRIAL: NCT01391897
Title: Epigenetics of Posttraumatic Stress Disorder and Somatoform Disorders in the Course of Psychotherapy
Acronym: TREPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Stefan Martin Henniger, MD., Department of Psychosomatic Medicin and Psychotherapy, Hannover Medical School, Hannover, Germany
Other Study IDs: MHH-EK-5689
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-06

CONDITIONS: Psychiatric Disorder; Somatoform Disorders; PTSD
Keywords: somatoform disorders; PTSD; epigenetics; psychotherapy; psychosomatics
MeSH Terms: conditions — Mental Disorders; Somatoform Disorders; Stress Disorders, Post-Traumatic | interventions — Psychotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- in- and out-patient psychotherapy patients: All included patients are highly selected in- and outpatients in a department of psychosomatic medicine (Germany) undergoing high dose psychotherapy (e.g. group therapy, creative therapy, cbt and psychodynamic psychotherapy).
  Interventions: Behavioral: psychotherapy

INTERVENTIONS:
Behavioral: psychotherapy — "multimodal complex psychotherapy"
  Other Names: all patients in the department are primarily included. There are no parallel groups.

SUMMARY:
This reported observational clinical study aims at identifying epigenetic markers in a sample of patients undergoing high dose inpatient psychotherapy suffering from a variety of psychiatric/psychosomatic diseases such as somatoform disorders, posttraumatic stress disorder (PTSD), depression, anxiety disorders and eating disorders.

The exact epigenetic markers that will be traced are yet to define.

The investigators believe that

1. Epigenetic patterns found in the group of psychiatric patients show differences from healthy controls
2. Different diagnosis show differences in epigenetic patterns as well
3. Epigenetic patterns correlate to the severity of the psychosocial disorder as measured in interviews or psychometric ratings
4. Epigenetic patterns can change under inpatient high dose psychotherapy
5. Changes correlate to clinical psychometric variables.

ELIGIBILITY:
Inclusion Criteria:

* informed consent given by the patient
* adulthood to 65 years
* stabel physical health
* at least fluent in German language (as it is a group-therapy)

Exclusion Criteria:

* psychiatric disorder such as substance addiction, psychosis, schizophrenia.
* insufficient understanding of the terms and conditions of the study
* insufficient emotional stability to fill out the psychometric forms required for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The present study includes all patients selected for multi-modal inpatient or day-clinic treatment in the department of psychosomatic medicine (as part of the centre of psychiatry)of the hannover medical school - given the informed consent of the patients. The patients treated in this unit are first seen in primary care and sent to us because of e.g. depression, somatization, eating-disorders, panic disorders, PTSD, or other psychiatric diseases commonly refered to as "psychosomatic" in Germany. They are subject to at least 2 diagnostic sessions in which further treamtment options are assessed.
  For about one third of the patients with grave psychiatric disorders, intensive "multimodal" psychotherapy in an inpatient or day-clinic setting is recommended.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-09 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- HannoverMS, Hanover, Lower Saxony, Germany